CLINICAL TRIAL: NCT06420193
Title: Evaluating the Feasibility and Acceptability of Study Procedures for a Full Factorial Trial of the AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
Brief Title: Evaluating Procedures for a Study of the AYA Survivors Coping and Emotional Needs Toolkit
Acronym: ASCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karly M Murphy, PhD, Principal Investigator, East Carolina University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-001795; R00CA248701 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Depression; Cancer; Adolescent; Young Adult; Adult
MeSH Terms: conditions — Depression; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Condition 1 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 2 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 3 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 4 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 5 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 6 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 7 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 8 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness)
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 9 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 10 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 11 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 12 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 13 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 14 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 15 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance)
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 16 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); and Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness)
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)

INTERVENTIONS:
Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT) — Participants will receive access to a digital depression self-management tool (ASCENT), which aims to help AYAs manage symptoms of depression post-treatment. All users will have access to the core tool which includes daily mood tracking and a psychoeducational module about cancer and depression. Depending on assigned condition, participants will also receive access to up to 4 intervention modules which have been adapted from existing evidence-based treatments for digital delivery to AYAs through a rigorous user-centered design process. Within each module there are 6 micro-lessons that include an educational video, a real story from an AYA that demonstrates the topic, multiple choice questions that ask the participant to apply the educational information to the AYA story, open-ended questions that ask the participant to apply the educational information to their own experience, and a practice activity in which they are asked to try out a relevant skill.

SUMMARY:
The investigators developed a digital intervention that aims to help adolescent and young adult cancer survivors (AYAs) manage symptoms of depression. This tool includes daily mood tracking, a psychoeducational module about cancer and depression, four components that are based on evidence-based interventions for depression. The goal of this study is to evaluate the acceptability of procedures for a future trial in which the investigators will test which component or combination of components meaningfully contribute to improvements in depressive symptoms among AYAs. Additionally, the investigators will evaluate study feasibility as well as intervention acceptability, satisfaction, usability, and engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment (adolescents 15-17, emerging adults 18-25, young adults 26-39)
* Age at diagnosis (adolescents 12-17, emerging adults 15-25, young adults 15-39)
* Time since completion of treatment: 1 month to 5 years
* Language: Fluent in English (spoken and written)
* Technology: Own smart phone with data plan

Exclusion Criteria:

* Mental Health: Current diagnosis of severe or persistent mental illness
* Suicidality: Severe suicidal ideation (including plan and intent)

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Acceptability of Study Procedures - Quantitative | Week 6
  An investigator-developed survey will be used to evaluate acceptability of study procedures. Mean scale scores range from 1 to 4, with higher scores indicating greater acceptability. Descriptive statistics and exact 95% confidence intervals (CIs) will be calculated.
Acceptability of Study Procedures - Qualitative | Weeks 6-8
  An investigator-developed semi-structured interview will be used to evaluate acceptability of study procedures. Transcriptions of semi-structured interviews will undergo rapid qualitative analysis to characterize the reasons for sub-optimal acceptability of study procedures.

SECONDARY OUTCOMES:
Study Feasibility - Recruitment Rate | Upon enrollment of 16 participants
  Recruitment rate will be calculated as the number of participants enrolled in the study divided by the number of participants contacted.
Study Feasibility - Retention Rate | Week 6
  Retention will be defined as the proportion of patients who provide T1 (6 week) data. Patients who discontinue the intervention (refuse phone calls) but complete the outcome assessments will be counted in the numerator for calculating retention.
Intervention Acceptability - Quantitative | Week 6
  An investigator-developed survey will be used to evaluate acceptability of the intervention.
Intervention Satisfaction - Quantitative | Week 6
  An investigator-developed survey will be used to evaluate satisfaction with the intervention. Mean scale scores range from 1 to 4, with higher scores indicating greater satisfaction. Descriptive statistics and exact 95% confidence intervals (CIs) will be calculated.
Intervention Acceptability & Satisfaction - Qualitative | Weeks 6-8
  A semi-structured interview will be used to further characterize acceptability of and satisfaction with the intervention. Transcriptions of semi-structured interviews will undergo rapid qualitative analysis to characterize the reasons for sub-optimal acceptability of and satisfaction with the intervention.
System Usability Scale | Week 6
  The System Usability Scale (SUS) will be administered to evaluate perceived usability of ASCENT. SUS scores range from 0 to 100, with higher scores indicating greater usability. Descriptive statistics and exact 95% confidence intervals (CIs) will be calculated.
Intervention Adherence | Weeks 1-6
  Adherence will be calculated as the percentage of pages viewed by the participant within a module divided by the total number of pages in the module as indicated by metrics from the website. Mean adherence rate and exact 95% confidence intervals (CIs) for each intervention module will be calculated.
eHealth Engagement Scale | Week 6
  The eHealth Engagement Scale will be administered to evaluate how engaging users found ASCENT engagement. Mean scale scores range from 1 to 4, with lower scores indicating greater engagement. Descriptive statistics and exact 95% confidence intervals (CIs) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Karly M Murphy, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data collected from participants in this study will be preserved and shared in alignment with best practices for open science. Data will be submitted to Dataverse, a free NIH Generalist Repository Ecosystem Initiative (https://dataverse.org/researchers).
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Ingram KM, Glock R, Williamson L, Coffey A, Anctil R, Augustinovic A, Yang D, Victorson D, Schoemann AM, Liles D, Salsman JM. Evaluating the feasibility and acceptability of study procedures for a full factorial trial of ASCENT: protocol for a randomized pilot. Pilot Feasibility Stud. 2025 Nov 24;11(1):147. doi: 10.1186/s40814-025-01728-z. PMID 41287126